CLINICAL TRIAL: NCT03193047
Title: A Randomized, Double-Blind, Parallel Group, Multicenter Study to Evaluate the Efficacy and Safety of Bempedoic Acid (ETC-1002) 180mg QD When Added to Proprotein Convertase Subtilisin/Kexin Type 9 (PCSK9)-Inhibitor Therapy
Brief Title: Evaluation of the Efficacy and Safety of Bempedoic Acid (ETC-1002) 180mg When Added to PCSK9 Inhibitor Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Esperion Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1002-039
Record Dates: First submitted 2017-06-19; First posted 2017-06-20 (Actual); Results first posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-03

CONDITIONS: Hypercholesterolemia
Keywords: Cholesterol; PCSK9; Repatha; evolocumab; LDL-C
MeSH Terms: conditions — Hypercholesterolemia | interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid; evolocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- bempedoic acid (Experimental): Bempedoic acid 180mg tablet taken orally, once daily plus evolocumab (Repatha) 420mg injection once monthly
  Interventions: Drug: bempedoic acid 180mg; Drug: evolocumab
- placebo (Placebo Comparator): Matching placebo tablet taken orally, once daily plus evolocumab (Repatha) 420mg injection once monthly
  Interventions: Other: placebo; Drug: evolocumab

INTERVENTIONS:
Drug: bempedoic acid 180mg — Daily bempedoic acid 180mg tablet in addition to monthly PCSK9i (evolocumab) background therapy
  Other Names: ETC-1002
  Arms: bempedoic acid
Other: placebo — Daily matching placebo tablet in addition to monthly PCSK9i (evolocumab) background therapy
  Arms: placebo
Drug: evolocumab — Monthly PCSK9i (evolocumab) background therapy
  Other Names: Repatha

SUMMARY:
The purpose of this study is to determine if bempedoic acid (ETC-1002) 180mg added to PCSK9 inhibitor (evolocumab) therapy is effective and safe in patients with elevated LDL cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years or legal age of majority depending on regional law
* Fasting, calculated LDL-C at screening ≥160 mg/dL and following PCSK9i therapy ≥70 mg/dL
* Men and nonpregnant, nonlactating women

Exclusion Criteria:

* Heterozygous (HeFH) or Homozygous (HoFH) Familial Hypercholesterolemia
* Total fasting TG ≥500 mg/dL
* Renal dysfunction or a glomerulonephropathy; eGFR <30 mL/min/1.73 m2
* Known cardiovascular disease (CVD), peripheral arterial disease (PAD), or cerebrovascular disease (CD)
* History of type 1 or type 2 diabetes
* Uncontrolled hypertension
* Uncontrolled hypothyroidism
* Liver disease or dysfunction
* Gastrointestinal conditions or procedures (including Lap-Band® or gastric bypass)
* History of hematologic or coagulation disorders
* History of malignancy (except non-metastatic basal or squamous cell carcinoma of the skin and cervical carcinoma in situ)
* Unexplained creatine kinase (CK) >3 × ULN
* Use of a cholesterylester transfer protein (CETP) inhibitor in the last 12 months prior to screening, such as: anacetrapib, dalcetrapib, or evacetrapib
* Pregnant or breast feeding, or planning to become pregnant during treatment and/ or within 30 days after the end of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2018-01-29 (Actual); Study Completion 2018-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Haberman, MD, Study Director — Esperion Therapeutics, Inc.
Locations (1):
- L-MARC Research Center, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pinkosky SL, Newton RS, Day EA, Ford RJ, Lhotak S, Austin RC, Birch CM, Smith BK, Filippov S, Groot PHE, Steinberg GR, Lalwani ND. Liver-specific ATP-citrate lyase inhibition by bempedoic acid decreases LDL-C and attenuates atherosclerosis. Nat Commun. 2016 Nov 28;7:13457. doi: 10.1038/ncomms13457. PMID 27892461
- [Background] Stone NJ, Robinson JG, Lichtenstein AH, Bairey Merz CN, Blum CB, Eckel RH, Goldberg AC, Gordon D, Levy D, Lloyd-Jones DM, McBride P, Schwartz JS, Shero ST, Smith SC Jr, Watson K, Wilson PW, Eddleman KM, Jarrett NM, LaBresh K, Nevo L, Wnek J, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Smith SC Jr, Tomaselli GF; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2013 ACC/AHA guideline on the treatment of blood cholesterol to reduce atherosclerotic cardiovascular risk in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Jun 24;129(25 Suppl 2):S1-45. doi: 10.1161/01.cir.0000437738.63853.7a. Epub 2013 Nov 12. No abstract available. PMID 24222016
- [Background] Sharrett AR, Ballantyne CM, Coady SA, Heiss G, Sorlie PD, Catellier D, Patsch W; Atherosclerosis Risk in Communities Study Group. Coronary heart disease prediction from lipoprotein cholesterol levels, triglycerides, lipoprotein(a), apolipoproteins A-I and B, and HDL density subfractions: The Atherosclerosis Risk in Communities (ARIC) Study. Circulation. 2001 Sep 4;104(10):1108-13. doi: 10.1161/hc3501.095214. PMID 11535564
- [Background] Thompson PD, Clarkson P, Karas RH. Statin-associated myopathy. JAMA. 2003 Apr 2;289(13):1681-90. doi: 10.1001/jama.289.13.1681. PMID 12672737
- See also: World Health Organization Fact Sheet No. 317 — http://www.who.int/mediacentre/factsheets/fs317/en/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 170 participants were screened; out of 170, 59 participants were randomized. One participant never received study medication and withdrew from the study due to the Sponsor's decision.
Groups:
- Placebo Plus Evolocumab: Participants received a matching oral placebo tablet taken once a day, plus evolocumab 420 milligrams (mg) injected over 9 minutes once a month as background therapy.
- Bempedoic Acid Plus Evolocumab: Participants received a bempedoic acid 180 mg tablet orally once a day (with or without food), plus evolocumab 420 mg injected once a month over 9 minutes as background therapy.
Period: Overall Study
Arm/Group | Placebo Plus Evolocumab | Bempedoic Acid Plus Evolocumab
Started | 31 | 28
Completed | 29 | 28
Not Completed | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Participant Left State | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received at least 1 dose of study medication. Participants in this group were included in the treatment group that they received, regardless of their randomized treatment.
Groups:
- Bempedoic Acid Plus Evolocumab: Participants received a bempedoic acid 180 mg tablet orally once a day (with or without food), plus evolocumab 420 mg injected over 9 minutes once a month as background therapy.
- Total: Total of all reporting groups
Arm/Group | Placebo Plus Evolocumab | Bempedoic Acid Plus Evolocumab | Total
Number analyzed (Participants) | 30 | 28 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (11.16) | 62.0 (9.36) | 60.1 (10.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 21 | 36
  Male | 15 | 7 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 2 | 4 | 6
  White | 28 | 24 | 52
Baseline Low-Density Lipoprotein Cholesterol (L-DLC) Values [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] — Baseline LDL-C is defined as the average of the Month -1 (Screening Visit 4) and Day 1 values. If only 1 value was available, then that single value was used as Baseline.
  milligrams per deciliter (mg/dL) | 104.12 (32.121) | 102.09 (28.982) | 103.14 (30.395)
Baseline Total Cholesterol (TC) and Non-High-Density Lipoprotein Cholesterol (Non-HDL-C) Values [Mean (Standard Deviation); unit: mg/dL] — Baseline TC and non-HDL-C are defined as the average of the Month -1 (Screening Visit 4) and the Day 1 (Treatment Visit 1) values. If a missing value presented at Month -1 or Day 1, then the last non-missing value prior to the first dose of double-blind study medication (including unscheduled assessments) within Month -1 and Day 1 was used to compute the Baseline measurements.
  mg/dL
    TC | 190.33 (39.387) | 186.20 (38.343) | 188.34 (38.601)
    non-HDL-C | 132.95 (36.599) | 129.68 (36.301) | 131.37 (36.172)
Baseline Apolipoprotein B (apoB) Values [Mean (Standard Deviation); unit: mg/dL] — Baseline values are defined as the Day 1 value. If a missing value presented at Day 1, then the last non-missing value prior to the first dose of double-blind study medication (including unscheduled assessments) within Month -1 and Day 1 was used to compute the Baseline measurements. Population: Only those participants with data available were analyzed.
  mg/dL
    number analyzed (Participants) | 28 | 28 | 56
    (all) | 87.9 (23.80) | 87.5 (27.13) | 87.7 (25.29)
Baseline High-Sensitivity C-Reactive Protein (hs-CRP) Values [Median (Inter-Quartile Range); unit: milligrams per Liter] — Baseline values are defined as the Day 1 value. If a missing value presented at Day 1, then the last non-missing value prior to the first dose of double-blind study medication (including unscheduled assessments) within Month -1 and Day 1 was used to compute the Baseline measurements. Population: Only those participants with data available were analyzed.
  milligrams per Liter
    number analyzed (Participants) | 29 | 28 | 57
    (all) | 2.090 [1.120 to 4.690] | 3.125 [1.270 to 4.590] | 2.340 [1.170 to 4.640]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C) at Month 2
Description: Percent change from Baseline is calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value ) x 100. Baseline is defined as the average of the last two non-missing values within Month -1 (Screening Visit 4) and Day 1 (Treatment Visit 1) values (including unscheduled assessments). If only one value was available, then that single value was used at Baseline. Percent change from Baseline was analyzed using analysis of covariance (ANCOVA), with treatment group as a factor and Baseline as a covariate. Missing data were imputed using last observation carried forward (LOCF) (only post-Baseline values were carried forward).
Time Frame: Baseline; Month 2
Population: Modified Intent-to-Treat (mITT) Population: all randomized participants with a Baseline lipid value and at least 1 post-Baseline lipid value who received investigational medicinal product (IMP) within 2 days before the lipid measurement and evolocumab 420 mg within 30 days plus or minus 3 days before the lipid measurement
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Plus Evolocumab | Bempedoic Acid Plus Evolocumab
Number analyzed (Participants) | 26 | 27
percent change | 2.783 (3.412) | -27.478 (4.310)
Statistical Analysis 1: Comparison: Placebo Plus Evolocumab vs Bempedoic Acid Plus Evolocumab; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = -30.261, 95% CI 2-sided [-41.324 to -19.199], Standard Error of Mean 5.502 — (Bempedoic acid plus evolocumab) minus (placebo plus evolocumab)

2. Secondary Outcome: Percent Change From Baseline in LDL-C at Month 1
Description: Percent change from Baseline is calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value ) x 100. Baseline is defined as the average of the last two non-missing values within Month -1 (Screening Visit 4) and Day 1 (Treatment Visit 1) values (including unscheduled assessments). If only one value was available, then that single value was used at Baseline. Percent change from Baseline was analyzed using ANCOVA, with treatment group as a factor and Baseline as a covariate. Observed data were used for analysis.
Time Frame: Baseline; Month 1
Population: Modified Intent-to-Treat Population. Only those participants with data available were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Plus Evolocumab | Bempedoic Acid Plus Evolocumab
Number analyzed (Participants) | 25 | 26
percent change | 3.172 (2.700) | -32.712 (4.385)
Statistical Analysis 1: Comparison: Placebo Plus Evolocumab vs Bempedoic Acid Plus Evolocumab; Test type: Superiority; p < 0.001, ANCOVA; Lease squares mean difference = -35.884, 95% CI 2-sided [-46.303 to -25.466], Standard Error of Mean 5.159 — (Bempedoic acid plus evolocumab) minus (placebo plus evolocumab)

3. Secondary Outcome: Absolute Change From Baseline in LDL-C at Month 1 and Month 2
Description: Change from Baseline is calculated as the post-Baseline value minus the Baseline value. Baseline is defined as the average of the Screening Visit 4 and the Day 1 value. If only 1 value is available, then that single value is used as Baseline. Change from Baseline was analyzed using ANCOVA, with treatment group as a factor and Baseline as a covariate. Observed data were used for analysis at Month 1. Missing Month 2 data were handled by LOCF.
Time Frame: Baseline; Month 1 and Month 2
Population: Modified Intent-to-Treat Population. Only those participants with data available were analyzed.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | Placebo Plus Evolocumab | Bempedoic Acid Plus Evolocumab
Number analyzed (Participants) | 26 | 27
milligrams per deciliter (mg/dL)
  Month 1: number analyzed (Participants) | 25 | 26
  Month 1 | 1.75 (3.118) | -36.51 (46.41)
  Month 2 | -0.02 (3.386) | -29.92 (4.461)
Statistical Analysis 1: Comparison: Placebo Plus Evolocumab vs Bempedoic Acid Plus Evolocumab; Month 1; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = -38.25, 95% CI 2-sided [-49.558 to -26.944], Standard Error of Mean 5.602 — (Bempedoic acid plus evolocumab) minus (placebo plus evolocumab)
Statistical Analysis 2: Comparison: Placebo Plus Evolocumab vs Bempedoic Acid Plus Evolocumab; Month 2; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = -29.90, 95% CI 2-sided [-41.176 to -18.626], Standard Error of Mean 5.606 — (Bempedoic acid plus evolocumab) minus (placebo plus evolocumab)

4. Secondary Outcome: Percent Change From Baseline in Lipid Profile Parameters at Month 1 and Month 2
Description: Percent change from Baseline is calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value ) x 100. Baseline apolipoprotein B (apoB) is defined as the Day 1 value. Baseline total cholesterol (TC) and non-high-density lipoprotein cholesterol (non-HDL-C) are defined as the average of the Month -1 (Screening Visit 4) and the Day 1 (Treatment Visit 1) values. If a missing value presented at Month -1 or Day 1, then the last non-missing value prior to the first dose of double-blind study medication (including unscheduled assessments) within Month -1 and Day 1 was used to compute the Baseline measurements. Percent change from Baseline was analyzed using ANCOVA, with treatment group as a factor and Baseline as a covariate. Observed data were used for analysis at Month 1. Missing Month 2 data were handled by LOCF.
Time Frame: Baseline; Month 1 and Month 2
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Plus Evolocumab | Bempedoic Acid Plus Evolocumab
Number analyzed (Participants) | 26 | 27
percent change
  apo-B at Month 1: number analyzed (Participants) | 18 | 20
  apo-B at Month 1 | 0.547 (2.948) | -26.484 (4.175)
  non-HDL-C at Month 1: number analyzed (Participants) | 25 | 26
  non-HDL-C at Month 1 | 2.077 (2.378) | -29.563 (4.031)
  TC at Month 1: number analyzed (Participants) | 25 | 26
  TC at Month 1 | 1.170 (1.877) | -20.770 (3.025)
  apo-B at Month 2: number analyzed (Participants) | 24 | 26
  apo-B at Month 2 | 2.706 (2.182) | -21.763 (3.736)
  non-HDL-C at Month 2 | 1.285 (2.783) | -22.960 (3.951)
  TC at Month 2 | 0.557 (2.009) | -16.963 (3.228)
Statistical Analysis 1: Comparison: Placebo Plus Evolocumab vs Bempedoic Acid Plus Evolocumab; Apo B at Month 1; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = -27.031, 95% CI 2-sided [-37.509 to -16.553], Standard Error of Mean 5.150 — (Bempedoic acid plus evolocumab) minus (placebo plus evolocumab)
Statistical Analysis 2: Comparison: Placebo Plus Evolocumab vs Bempedoic Acid Plus Evolocumab; Apo B at Month 2; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = -24.469, 95% CI 2-sided [-33.225 to -15.713], Standard Error of Mean 4.330 — (Bempedoic acid plus evolocumab) minus (placebo plus evolocumab)
Statistical Analysis 3: Comparison: Placebo Plus Evolocumab vs Bempedoic Acid Plus Evolocumab; non-HDL-C at Month 1; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = -31.640, 95% CI 2-sided [-41.116 to -22.163], Standard Error of Mean 4.689 — (Bempedoic acid plus evolocumab) minus (placebo plus evolocumab)
Statistical Analysis 4: Comparison: Placebo Plus Evolocumab vs Bempedoic Acid Plus Evolocumab; non-HDL-C at Month 2; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = -24.246, 95% CI 2-sided [-33.987 to -14.505], Standard Error of Mean 4.838 — (Bempedoic acid plus evolocumab) minus (placebo plus evolocumab)
Statistical Analysis 5: Comparison: Placebo Plus Evolocumab vs Bempedoic Acid Plus Evolocumab; TC at Month 1; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = -21.941, 95% CI 2-sided [-29.153 to -14.729], Standard Error of Mean 3.572 — (Bempedoic acid plus evolocumab) minus (placebo plus evolocumab)
Statistical Analysis 6: Comparison: Placebo Plus Evolocumab vs Bempedoic Acid Plus Evolocumab; TC at Month 2; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = -17.520, 95% CI 2-sided [-25.201 to -9.839], Standard Error of Mean 3.809 — (Bempedoic acid plus evolocumab) minus (placebo plus evolocumab)

5. Secondary Outcome: Percent Change From Baseline in High-sensitivity C-reactive Protein (Hs-CRP) at Month 1 and Month 2
Description: Percent change from Baseline is calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value ) x 100. Baseline is defined as the Day 1 value. Percent change from Baseline was analyzed using a non-parametric approach. Missing Month 2 data were handled by LOCF. Observed data were used for analysis at Month 1.
Time Frame: Baseline; Month 1 and Month 2
Population: Modified Intent-to-Treat Population. Only those participants with data available were analyzed.
Measure: Median (Inter-Quartile Range); unit: percent change
Groups:
- Placebo + Evolocumab: Participants received matching oral placebo tablet taken once a day, plus evolocumab 420 milligrams (mg) injected over 9 minutes once a month as background therapy.
- Bempedoic Acid + Evolocumab: Participants received oral bempedoic acid 180 mg tablet once a day (with or without food), plus evolocumab 420 mg injected once a month over 9 minutes as background therapy.
Arm/Group | Placebo + Evolocumab | Bempedoic Acid + Evolocumab
Number analyzed (Participants) | 26 | 27
percent change
  hs-CRP at Month 1: number analyzed (Participants) | 24 | 26
  hs-CRP at Month 1 | 10.658 [-36.488 to 66.374] | -23.349 [-57.857 to 5.128]
  hs-CRP at Month 2: number analyzed (Participants) | 25 | 27
  hs-CRP at Month 2 | -1.623 [-39.445 to 26.531] | -34.444 [-57.599 to -7.083]
Statistical Analysis 1: Comparison: Placebo + Evolocumab vs Bempedoic Acid + Evolocumab; hs-CRP at Month 1; Test type: Superiority; p = 0.046, Wilcoxon rank sum test; Median treatment difference = -32.479, 95% CI 2-sided [-70.524 to -2.339], Standard Error of Mean 17.395 — The median treatment difference (location shift) and the 95% confidence limits are from Hodges-Lehmann estimates
Statistical Analysis 2: Comparison: Placebo + Evolocumab vs Bempedoic Acid + Evolocumab; hs-CRP at Month 2; Test type: Superiority; p = 0.029, Wilcoxon rank sum test; Median treatment difference = -28.512, 95% CI 2-sided [-51.455 to -3.930], Standard Error of Mean 12.124 — The median treatment difference (location shift) and the 95% confidence limits are from Hodges-Lehmann estimates

6. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (AE) and Treatment-emergent Serious Adverse Event (SAE)
Description: Treatment-emergent AEs (TEAEs) and SAEs (TESAEs) were reported and defined as any AE that began or worsened after the first dose of investigational medicinal product.
Time Frame: up to Month 2 (until 30 days after last dose)
Population: Safety Population: all randomized participants who received at least 1 dose of IMP. Participants in the Safety Population were included in the treatment group that they received, regardless of their randomized treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Evolocumab | Bempedoic Acid + Evolocumab
Number analyzed (Participants) | 30 | 28
Participants
  Any TEAE | 7 | 9
  TEAEs related to IMP | 1 | 1
  TEAEs related to evolocumab | 1 | 0
  TESAEs | 0 | 1
  TESAEs related to IMP | 0 | 0
  TESAEs related to evolocumab | 0 | 0
  Deaths | 0 | 0
  Discontinuation of IMP due to TEAE | 0 | 0
  Mild TEAEs | 5 | 4
  Moderate TEAEs | 2 | 4
  Severe TEAEs | 0 | 1

7. Secondary Outcome: Number of Participants With Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) >3x the Upper Limit of Normal (ULN) at Month 1 and Month 2
Description: The number of participants with ALT or AST >3x ULN was measured.
Time Frame: Month 1 and Month 2
Population: Safety Population. Only those participants with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Plus Evolocumab | Bempedoic Acid Plus Evolocumab
Number analyzed (Participants) | 30 | 28
Participants
  ALT, Month 1: number analyzed (Participants) | 28 | 27
  ALT, Month 1 | 0 | 0
  ALT, Month 2: number analyzed (Participants) | 29 | 28
  ALT, Month 2 | 0 | 0
  AST, Month 1: number analyzed (Participants) | 28 | 28
  AST, Month 1 | 0 | 0
  AST, Month 2: number analyzed (Participants) | 28 | 28
  AST, Month 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: up to Month 2 (until 30 days after last dose)
Description: Treatment-emergent adverse events (TEAEs) and serious TEAEs, defined as those events that began or worsened after the first dose of investigational medicinal product (IMP) until 30 days after the last dose of IMP, were reported for the Safety Population.
Arm/Group | Placebo Plus Evolocumab | Bempedoic Acid Plus Evolocumab
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/30 | 1/28
Other Adverse Events (participants affected / at risk) | 7/30 | 8/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Plus Evolocumab (N=30) | Bempedoic Acid Plus Evolocumab (N=28)
Influenza (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Plus Evolocumab (N=30) | Bempedoic Acid Plus Evolocumab (N=28)
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Injection site reaction (General disorders) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Ejaculation failure (Reproductive system and breast disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If the Principal Investigator plans to publish information from the study, a copy of the manuscript should be provided to the Sponsor for review before submission for publication or presentation. The Sponsor may request that that publication be withheld.

DOCUMENTS (2):
  • Study Protocol (2017-03-05): https://cdn.clinicaltrials.gov/large-docs/47/NCT03193047/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT03193047/SAP_001.pdf